CLINICAL TRIAL: NCT02419742
Title: An Indian Multicentric Open Label Prospective Phase IV Study to Evaluate Safety and Efficacy of Trastuzumab in Her2 Positive, Node Positive or High Risk Node Negative Breast Cancer as Part of a Treatment Regimen Consisting of Doxorubicin, Cyclophosphamide, With Either Docetaxel or Paclitaxel (AC-TH) or Docetaxel and Carboplatin (TCH)
Brief Title: Safety and Efficacy of Trastuzumab as Part of Breast Cancer Treatment Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28714
Record Dates: First submitted 2015-03-23; First posted 2015-04-17 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Cyclophosphamide; Docetaxel; Doxorubicin; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trastuzumab (Experimental): Participants will receive trastuzumab as a part of either AC-TH or TCH treatment regimen. The choice of the regimen will be based on investigator's discretion referring the local prescribing document of trastuzumab. AC-TH consists of doxorubicin and cyclophosphamide followed by either paclitaxel or docetaxel. TCH consists of docetaxel and carboplatin. Trastuzumab will be common in both treatment regimens and could be administered weekly or every 3 weeks, as per investigator discretion. Each cycle will be of 3 weeks.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Carboplatin — TCH regimen: Carboplatin dose = Target Area Under Curve (AUC) (6 milligrams*milliliter/minute [mg*mL/min]) multiplied by (Glomerular Filtration Rate [GFR] + 25). Carboplatin will be administered as IV bolus every 3 weeks for 6 cycles (Cycles 1 to 6).
Drug: Cyclophosphamide — AC-TH regimen: Cyclophosphamide 600 mg/m^2 IV bolus every 3 weeks for 4 cycles (Cycles 1 to 4).
Drug: Docetaxel — AC-TH regimen: Docetaxel 100 mg/m^2 IV infusion every 3 weeks for 4 cycles (Cycles 5 to 8). TCH regimen: Docetaxel 75 mg/m^2 IV bolus every 3 weeks for 6 cycles (Cycles 1 to 6).
Drug: Doxorubicin — Participants will receive Doxorubicin 60 mg/m^2 administered as I.V. bolus injection over 5 to 15 minute every 3 weeks for 4 cycles for AC-TH regimen.
Drug: Paclitaxel — AC-TH regimen: Paclitaxel 175 mg/m^2 IV infusion every 3 weeks for 4 cycles (Cycles 5 to 8).
Drug: Trastuzumab — AC-TH regimen: For weekly administration, 4 milligrams per kilograms (mg/kg) loading dose on Day 1 of Cycle 5, followed by 2 mg/kg on Day 8 of Cycle 5 and 2 mg/kg every week for 4 cycles (up to Cycle 8). For 3 weekly administration, 8 mg/kg loading dose on Day 1 of Cycle 5, followed by 6 mg/kg every 3 for 4 cycles (up to Cycle 8). From Day 1 of Cycle 9, 6 mg/kg will be administered every 3 weeks up to Cycle 22. TCH regimen: For weekly administration, 4 mg/kg loading dose followed by 2 mg/kg weekly from Cycles 1 to Cycle 6. For 3 weekly administration, 8 mg/kg loading dose followed 6 mg/kg every 3 weeks from Cycles 1 to 6. From Cycle 7, 6 mg/kg every 3 weeks up to Cycle 18. All administrations will be intravenous (IV) infusion.

SUMMARY:
This is a prospective, Phase IV, multi-center, single arm, open-label, interventional study to evaluate the safety of trastuzumab for the treatment of human epidermal growth factor receptor 2 protein (HER2)-positive node positive or high risk node negative breast cancer participants with regimen consisting of doxorubicin and cyclophosphamide followed by either paclitaxel or docetaxel (AC-TH Regimen) or a regimen consisting of docetaxel and carboplatin (TCH Regimen) in Indian population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed early invasive HER2 positive, node positive or high risk node negative breast cancer with no evidence of residual, locally recurrent or metastatic disease and defined as clinical stage I to IIIA that is eligible for adjuvant treatment with trastuzumab
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* HER2 over expression/amplification defined as either Immunohistochemistry (IHC)3+, or IHC2+ and Fluorescence in situ Hybridization (FISH) positive as determined in a central laboratory
* At time of starting trastuzumab therapy, LVEF measured by echocardiography
* Screening LVEF greater than or equal to (>/=) 55 percent (%)
* Adequate bone marrow, renal, and hepatic function
* Agreement to use an adequate, non-hormonal means of contraception by women of childbearing potential

Exclusion Criteria:

* Any contraindication to trastuzumab
* Previous adjuvant breast cancer treatment with an approved or investigational anti-HER2 agent
* History of other malignancy, except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma and participants with other curatively treated malignancies who have been disease-free for at least 5 years
* Past history of ductal carcinoma in situ and/or lobular carcinoma that has been treated with any systemic therapy or with radiation therapy to the ipsilateral breast where the invasive cancer subsequently develops
* Locally advanced (Stage IIIB and IIIC) and metastatic disease (Stage IV)
* Clinically relevant cardiovascular disorder or disease
* Uncontrolled hypertension, or history of hypertensive crisis or hypertensive encephalopathy
* History of severe allergic or immunological reactions, example difficult to control asthma
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kukreja, MD, Study Director — Roche Products (India) Pvt. Ltd.
Locations (6):
- India (6):
  - Yashoda Hospital, Hyderabad, Andhra Pradesh
  - Manipal Hospital; Department of Oncology, Bangalore, Karnataka
  - Jehangir Clinical Development Centre Pvt. Ltd; Cancer Research Room, Pune, Maharashtra
  - Rajiv Gandhi Cancer Institute & Research Center, New Delhi, National Capital Territory of Delhi
  - MAX Balaji Hospital, Delhi
  - Dr. GVN Cancer Institute; Medical Oncology, Trichy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 investigational sites in India.
Pre-assignment Details: Of the 110 participants enrolled, 108 received at least one dose of trastuzumab and were included in the safety population.
Groups:
- Trastuzumab With AC-TH Regimen: Participants received trastuzumab with AC-TH regimen. The choice of the regimen was based on the investigator's discretion referring the local prescribing document of trastuzumab. AC-TH regimen consisted of doxorubicin and cyclophosphamide followed by either paclitaxel or docetaxel. Trastuzumab was common in both treatment regimens and was administered weekly or every 3 weeks, as per investigator discretion. Each cycle was 3 weeks.
- Trastuzumab With TCH Regimen: Participants received trastuzumab with TCH regimen. The choice of the regimen was based on the investigator's discretion referring the local prescribing document of trastuzumab. TCH consisted of docetaxel and carboplatin. Trastuzumab was common in both treatment regimens and was administered weekly or every 3 weeks, as per investigator discretion. Each cycle was 3 weeks.
Period: Overall Study
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
Started | 58 | 52
Completed | 53 | 50
Not Completed | 5 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Disease Progression | 0 | 1
Not completed — Withdrew Consent | 2 | 1
Not completed — Any other reason which the Investigator deemed participant unsuitable for enrollment into the study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen | Total
Number analyzed (Participants) | 58 | 52 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.95 (7.96) | 51.19 (10.94) | 51.59 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 52 | 110
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 58 | 52 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Changes in Cardiac Function As Determined by Left Ventricular Ejection Fraction (LVEF) Measurements Using Echocardiography
Description: LVEF assessments were performed every three months (four cycles) using echocardiogram
Time Frame: Baseline to every 4 cycles up to Cycle 21 (AC-TH), every 4 cycles up to Cycle 17 (TCH) (each cycle is 21 days), at study treatment completion (12 months post baseline) at 6 month (18 months post baseline) and 12 month follow-up (24 months post baseline)
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
Number analyzed (Participants) | 56 | 52
Percentage of LVEF
  Baseline | 60.1 (6.17) | 62.1 (2.30)
  Cycle 5: number analyzed (Participants) | 56 | 49
  Cycle 5 | -0.2 (4.71) | -0.4 (2.72)
  Cycle 9: number analyzed (Participants) | 54 | 47
  Cycle 9 | -0.5 (4.64) | -1.0 (2.98)
  Cycle 13: number analyzed (Participants) | 53 | 49
  Cycle 13 | -2.0 (6.94) | -1.0 (2.36)
  Cycle 17: number analyzed (Participants) | 54 | 49
  Cycle 17 | -1.8 (4.77) | -1.1 (3.15)
  Cycle 21: number analyzed (Participants) | 52 | 0
  Cycle 21 | -1.8 (4.88) |
  Study Completion Visit: number analyzed (Participants) | 56 | 48
  Study Completion Visit | -3.3 (6.59) | -0.7 (2.72)
  6 Month Follow Up: number analyzed (Participants) | 38 | 44
  6 Month Follow Up | -1.6 (5.89) | -0.3 (3.18)
  12 Month Follow Up: number analyzed (Participants) | 30 | 46
  12 Month Follow Up | -2.2 (6.28) | -0.4 (2.92)

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the treatment. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study were also considered as adverse events.
Time Frame: Baseline up to approximately 5 years and 10 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
Number analyzed (Participants) | 56 | 52
Participants | 46 | 51

3. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS was defined as time from the date of first study treatment to the date of local, regional or distant recurrence, contra-lateral breast cancer or death due to any cause. Local, regional or distant recurrence, and contra-lateral breast cancer was assessed by combination of physical examination, mammography and pelvic examination.
Time Frame: The date of first study treatment to the date of local, regional or distant recurrence, contra-lateral breast cancer or death due to any cause within 12 months from the last dose of Trastuzumab for every participant
Population: ITT population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
Number analyzed (Participants) | 58 | 52
Months | NA [NA to NA] — The median duration of DFS was not estimable as there were no disease progression during the study period. | NA [NA to NA] — The median duration of DFS was not estimable as there were no disease progression during the study period.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as time from the date of first study treatment until date of death, regardless of the cause of death.
Time Frame: Time from the date of first study treatment until date of death, regardless of the cause of death within 12 months from the last dose of Trastuzumab for every participant. The follow up period was 52 weeks from the last dose of treatment in both arms.
Population: ITT population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
Number analyzed (Participants) | 58 | 52
Months | NA [NA to NA] — The median duration of OS was not estimable because no deaths were reported during the study. The deaths occurred during the monitoring period of adverse events for the overall study, but not during the overall survival time frame and were censored for OS analysis. | NA [NA to NA] — The median duration of OS was not estimable because no deaths were reported during the study. The deaths occurred during the monitoring period of adverse events for the overall study, but not during the overall survival time frame and were censored for OS analysis.

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 5 years and 10 months
Arm/Group | Trastuzumab With AC-TH Regimen | Trastuzumab With TCH Regimen
All-Cause Mortality (participants affected / at risk) | 1/56 | 1/52
Serious Adverse Events (participants affected / at risk) | 11/56 | 9/52
Other Adverse Events (participants affected / at risk) | 46/56 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab With AC-TH Regimen (N=56) | Trastuzumab With TCH Regimen (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab With AC-TH Regimen (N=56) | Trastuzumab With TCH Regimen (N=52)
Leukopenia (Blood and lymphatic system disorders) | 22 (56) | 3 (3)
Urinary tract infection (Infections and infestations) | 14 (23) | 3 (3)
Pyrexia (General disorders) | 12 (18) | 11 (15)
Anaemia (Blood and lymphatic system disorders) | 12 (19) | 27 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 3 (5)
Peripheral motor neuropathy (Nervous system disorders) | 6 (7) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 4 (9)
Ejection fraction decreased (Investigations) | 5 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 9 (11)
Fatigue (General disorders) | 3 (3) | 8 (11)
Pain (General disorders) | 3 (4) | 3 (5)
Paronychia (Infections and infestations) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (11)
Paraesthesia (Nervous system disorders) | 3 (3) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 22 (30)
Asthenia (General disorders) | 0 (0) | 12 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (11)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 8 (13)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
Headache (Nervous system disorders) | 0 (0) | 7 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 6 (7)
Peripheral swelling (General disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 4 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2013-07-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02419742/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT02419742/SAP_001.pdf